CLINICAL TRIAL: NCT06824662
Title: A Phase 0/1b 'Trigger' Clinical Trial With an Expansion Phase of Quisinostat Plus Fractionated Radiotherapy in Newly-diagnosed and Recurrent Grade 4 IDH-WT Glioblastomas
Brief Title: Phase 0 With Expansion Phase Clinical Trial of Quisinostat Plus Radiotherapy in Newly-diagnosed and Recurrent Grade 4 IDH-Wildtype Glioblastomas
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Responsible Party: Sponsor-Investigator, Nader Sanai, Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-18
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma WHO Grade IV
Keywords: IDH-WT
MeSH Terms: interventions — quisinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Recurrent WHO Grade 4 Glioblastoma IDH-WT (Experimental)
  Interventions: Drug: Quisinostat
- Newly-Diagnosed WHO Grade 4 Glioblastoma IDH-WT (Experimental)
  Interventions: Drug: Quisinostat

INTERVENTIONS:
Drug: Quisinostat — a highly potent and orally active HDAC inhibitor

SUMMARY:
This is an open-label, multi-center Phase 0/1b study that will enroll up to 18 participants with recurrent WHO grade 4 glioblastoma (rGBM) IDH-wildtype (IDH-WT), Arm A, and 12 participants with presumed newly-diagnosed WHO grade 4 glioblastoma (nGBM) IDH-WT, Arm B. The trial will be composed of a Phase 0 component (subdivided into Arms A and B), and an Expansion Phase 1b. Patients with tumors demonstrating a positive pharmacokinetic (PK) response in the Phase 0 component of the study will graduate to an Expansion Phase that combines therapeutic dosing of quisinostat plus standard-of-care fractionated radiotherapy (RT).

DETAILED DESCRIPTION:
Eligible participants (rGBM in Arm A and nGBM in Arm B) will enroll in the Phase 0 study and receive quisinostat prior to a planned resection. Arm A includes a 3+3 design to determine optimal time interval (OTI) of final dose prior to surgery. Further rGBM participants and nGBM participants will enroll at OTI once established. Blood, tumor, and cerebrospinal fluid (CSF) samples will be collected during surgery, and blood and CSF samples will be collected after surgery, to measure the amount of drug that is present in the samples. Participants with tumors demonstrating PK response will continue with therapeutic dosing of quisinostat treatment on Monday, Wednesday, Friday of 5-day cycles after surgery concurrently with their standard of care (SOC) fractionated RT. Participants will continue to receive quisinostat and SOC RT for their physician-directed duration of RT, (2-3 weeks for rGBM and 5-6 weeks form nGBM).

The Phase 0 Primary Objective is to evaluate concentration of quisinostat in gadolinium-non-enhancing tumor tissue, and the Expansion Phase Primary Objective is to determine the 6-month progression free survival (PFS6) rate in rGBM participants who had positive PK response in Phase 0.

The Phase 0 Secondary Objective is to evaluate concentration of quisinostat in CSF, and the Expansion Phase Secondary Objectives are to monitor safety and tolerability of quisinostat and examine overall survival (OS) in participants.

ELIGIBILITY:
Inclusion Criteria:

* For Arm A: Participants who have had a prior resection of diagnosed glioblastoma, IDH wildtype (2021 WHO grade 4), defined as participants who have progressed on or following standard therapy, which includes maximal surgical resection, temozolomide, and fractionated radiotherapy. Participants will also need to have radiation planned as part of the post-surgical treatment plan; OR, for Arm B only: Participants undergoing resection for a suspected newly diagnosed WHO Grade 4 glioblastoma, IDH wildtype. Participants will also need to have radiation planned as part of the post-surgical treatment plan.
* Participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm.
* Provision of signed and dated, written informed consent (personally or by the legally authorized representative, if applicable) prior to any study specific procedures, sampling and analyses.
* Age ≥18 at time of consent
* Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Ability to swallow oral medications.
* Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):
* Participants with tumor-induced seizures must be well-controlled on a stable anti-epileptic treatment.
* Participants must be willing to receive prophylaxis with levetiracetam for the duration of study drug administration (or alternative anti-epileptic if agreed with Medical Monitor).
* Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
* For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation until the end of treatment administration and for 16 weeks after the last dose of study drug.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner until the end of treatment administration and for 16 weeks after the last dose of study drug.
* Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

* Pregnancy or lactation.
* Known allergic reactions to components of the quisinostat.
* Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis, as determined by the investigator.
* Known active systemic bacterial infection (requiring intravenous [IV] antibiotics or fever >38.5°C at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening of viral infection is not required for enrollment.
* The participant has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Any of the following cardiac criteria: cardiac dysfunction defined as myocardial infarction within six months of study entry, NYHA Class II/III/IV heart failure, unstable angina or unstable cardiac arrhythmias; mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs) (QTc interval will be calculated using Fridericia's formula); any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block; any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age (patients stable on concomitant medications known to prolong the QT interval may be allowed to participate in the study provided that their mean resting corrected QT interval (QTcF) is < 450 msec in males or < 470msec in females at baseline and after discussion with the Principal Investigator); use of medications that may cause Torsades de Pointes.
* History or presence of myopathy or raised creatine kinase (CK) > 5 x upper limit of normal (ULN) on 2 occasions at screening.
* Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30 ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Prior therapy with histone-deacetylase inhibitor therapy; more than 3 prior lines of therapy.
* Treatment with strong inhibitors or inducers of CYP3A4 within 2 weeks prior to receiving study drug.
* Prior treatment with pneumotoxic drugs, e.g. busulfan, bleomycin, within the past year. If prior therapy in lifetime, then excluded if history of pulmonary toxicities from administration. Patients who have received treatment with nitrosoureas (e.g., BCNU, CCNU) in the year before study entry without experiencing lung toxicity are allowed on study.
* Treatment with another investigational drug or other intervention within 5 half-lives of the investigational product, whichever is longer.
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) Grade 1 at the time of starting study treatment and patients with chronic Grade 2 unresolved toxicities may be eligible following discussion with the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Quisinostat Concentration in Tumor Tissue | Phase 0 surgery
  Total and unbound quisinostat concentration will be quantified in Gd-enhancing and Gd-non-enhancing tumor tissue collected during Phase 0 surgery.
6-Month Progression Free Survival (PFS6) Rate in Participants | From date of Phase 0 surgery to date of disease recurrence or death, assessed over 16 months
  The rate of 6-month progression-free survival of participants that had a positive PK response (defined as unbound concentrations of quisinostat equal or greater than 0.5 nM in Gd-non-enhancing tumor tissue) will be quantified.

SECONDARY OUTCOMES:
Quisinostat Concentration in Cerebrospinal Fluid (CSF) | From date of Phase 0 surgery through study completion, assessed over 4 months
  Quisinostat concentration will be quantified in cerebrospinal fluid collected during Phase 0 surgery and throughout study duration of participants with an Ommaya reservoir and shunt placed during surgery.
Number of Participants with Drug-Related Toxicity | From date of first dose until 30 days after last dose, assessed over 4 months
  Safety and tolerability of quisinostat will be assessed by tabulating the number of drug-related toxicities (graded per CTCAE version 5) which include:
  * Grade 2 or higher cardiac disorder
  * Grade 4 or higher hematological or nonhematological toxicity
  * Febrile neutropenia
  * Unacceptable toxicity as determined by the Investigator
  * Any Grade 3 or higher non-hematologic toxicity, excluding the following: Grade 3 nausea, vomiting, or diarrhea for less than 72 hours with adequate supportive care; Grade 3 fatigue for longer than 1 week; Grade 3 or higher electrolyte abnormality lasting up to 72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional treatment
Number of Treatment-Emergent Adverse Events | From date of enrollment until 30 days after last dose, assessed over 6 months
  Safety and tolerability of quisinostat will be assessed by tabulating participants that had treatment-emergent adverse events according to the highest Grade observed per patient for each event or category (graded per CTCAE version 5).
Number of Treatment-Related Adverse Events | From date of first dose until 30 days after last dose, assessed over 4 months
  Safety and tolerability of quisinostat will be assessed by tabulating participants that had treatment-related adverse events (defined as those events definitely, probably, or potentially related to study treatment) according to the highest Grade observed per patient for each event or category (graded per CTCAE version 5).
Number of Participants with Clinical Laboratory Abnormalities | From date of first dose until 30 days after last dose, assessed over 4 months
  Safety and tolerability of quisinostat will be assessed by tabulating participants that had clinical laboratory abnormalities stratified by each event or abnormal result.
Number of Serious Adverse Events and Deaths | From date of enrollment until 30 days after last dose, assessed over 6 months
  Safety and tolerability of quisinostat will be assessed by aggregating and tabulating participants that died during study participation (due to any cause), and participants that had serious adverse events according to the highest Grade observed per patient for each event or category (graded per CTCAE version 5).
Overall Survival during Expansion Phase | From date of surgery until death, assessed up to 16 months
  Overall Survival of participants that had a positive PK response (defined as unbound concentrations of quisinostat equal or greater than 0.5 nM in Gd-non-enhancing tumor tissue) will be summarized using Kaplan-Meier Curves and Estimates.

OTHER OUTCOMES:
Systemic PK: Peak Plasma Concentration (Cmax) | From date of first dose until standard of care post-op follow-up visit, assessed over 1 month
  Peak plasma concentration (Cmax) of total and unbound quisinostat levels will be quantified.
Systemic PK: Time to Peak Plasma Concentration (Tmax) | From date of first dose until standard of care post-op follow-up visit, assessed over 1 month
  Time to peak plasma concentration (Tmax) of total and unbound quisinostat levels will be quantified.
Systemic PK: Quisinostat Half-Life (T1/2) in Plasma | From date of first dose until standard of care post-op follow-up visit, assessed over 1 month
  The half-life (T1/2) of total and unbound quisinostat levels in plasma will be quantified.
Systemic PK: Area Under Time/Concentration Curve (AUC0-24) in Plasma | From time of last dose assessed over 24 hours
  Area under the time/concentration curve (AUC0-24) over 24 hours of total and unbound quisinostat levels in plasma will be quantified.
Total (Kp) and Unbound (Kp,uu) Partition Coefficient of Quisinostat | From date of first dose to 30 days after last Phase 0 dose, assessed over 2 months
  The tumor to plasma partition coefficients of quisinostat for total (Kp) and unbound (Kp,uu) drug levels will be quantified.
Change in Biomarker Concentrations in Tumor Tissue | Baseline, Phase 0 surgery
  Tumor tissue collected during surgery will be compared to baseline tissue to assess fold induction change of AcH3K9/14, pH2AX, ClCas-3, and MIB-1.
Changes in Cell State and Gene Expression of Tumor Tissue | Phase 0 surgery, subsequent surgery(ies)
  Tumor tissue collected at subsequent resections (if any) will be compared to tumor tissue collected during Phase 0 surgery to determine changes in cell state and gene expression using single-cell RNA-seq analysis.
Genomic Changes of DNA in CSF | Baseline, Phase 0 surgery, post-op follow-up, day 1 of each cycle assessed over 3 months
  Genomic changes will be assessed by sequencing DNA from tumor cells and/or cell-free DNA in CSF collected during Phase 0 surgery and throughout study duration of participants with an Ommaya reservoir and shunt placed during surgery.
Transcriptome Changes of RNA in CSF | Baseline, Phase 0 surgery, post-op follow-up, day 1 of each cycle assessed over 3 months
  Transcriptomic changes will be assessed by sequencing RNA from tumor cells in CSF collected during Phase 0 surgery and throughout study duration of participants with an Ommaya reservoir and shunt placed during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Ivy Brain Tumor Center
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No